CLINICAL TRIAL: NCT04349579
Title: Evaluation of the Effects of Irrigation of the Extraction Socket With Rifamycine on Postoperative Pain, Edema and Trismus in Impacted Lower Third Molar Surgery
Brief Title: Evaluation of the Effects of Irrigation of the Extraction Socket With Rifamycine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, levent Cigerim, Head of Oral and Maxillofacial Surgery Department, Yuzuncu Yil University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 19.07.2017/07
Record Dates: First submitted 2020-04-12; First posted 2020-04-16 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Impacted Third Molar Tooth
Keywords: rifamycine; pain; edema; trismus
MeSH Terms: conditions — Pain; Edema; Trismus | interventions — Rifamycins; Rifampin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifamycine (Experimental): Rifamycine is a broad spectrum semi-synthetic antibiotic that acts on gram-positive and gram-negative microorganisms. As a local application, it has areas of use in dentistry such as washing fistula mouths, maxillary sinus and abscess wounds and treating osteomyelitis.
  Interventions: Drug: Rifamycine
- Saline (Active Comparator): Saline, also known as saline solution, is a mixture of sodium chloride in water and has a number of uses in medicine. Applied to the affected area it is used to clean wounds. It is also used to dilute other drugs to be injected and to wash the operation site in dental surgery operations. It is most commonly used as a sterile 9 g of salt per litre (0.9%) solution, known as normal saline.
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Rifamycine — Local anesthesia was obtained using 2 ml articaine hydrochloride 40 mg/ml with epinephrine 0.01 mg/ml . The horizontal incision was made with no. 15 scalpel blade and a full thickness mucoperiosteal flap was raised. In all surgical procedures, bone removal and/or tooth sectioning were performed under sterile saline irrigation. Following the extraction, granulation tissues were removed, and bleeding was controlled. Finally, extraction socket was irrigated with the solution which contains 250 mg rifamycine and the mucoperiosteal flap was repositioned by 3.0 silk sutures.
  Other Names: RIF 250 MG IM Ampul
  Arms: Rifamycine
Drug: Saline Solution — Local anesthesia was obtained using 2 ml articaine hydrochloride 40 mg/ml with epinephrine 0.01 mg/ml . The horizontal incision was made with no. 15 scalpel blade and a full thickness mucoperiosteal flap was raised. In all surgical procedures, bone removal and/or tooth sectioning were performed under sterile saline irrigation. Following the extraction, granulation tissues were removed, and post extraction cavity was irrigated with saline solution. After the bleeding was controlled, the mucoperiosteal flap was repositioned by 3.0 silk sutures.
  Other Names: KANFLEKS % 0,9 IZOTONIK SODYUM KLORUR
  Arms: Saline

SUMMARY:
Removal of impacted lower third molar teeth is one of the most common oral surgical procedures, and these operations often lead to various complications in patients. Antibiotics, analgesics and mouthwashes are prescribed for the treatment of complications encountered. When using postoperative antibiotics in surgery of impacted third molar teeth, lower surgical area infection, pain, swelling and trismus are seen. Based on this information, in this study, it is aimed to evaluate the effects of rifamycine intraoperatively on the postoperative pain, swelling and trismus.

ELIGIBILITY:
Inclusion Criteria:

* absence of any systemic disease
* having bilateral impacted mandibular third molar teeth in a similar position
* absence of allergy to any of the drugs used in the study,
* absence of pregnancy/lactating state,
* no history of any medication use during at least 2 week before the operation.

Exclusion Criteria:

* not regularly coming to the controls,
* not using their medicines regularly
* using any additional medication that may affect the outcome of the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | Postoperatif 1st day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Pain | Postoperatif 2nd day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Swelling | Postoperative 2nd day
  Postoperative swelling was evaluated by the distance between predetermined facial anatomic landmarks (from the mandibular angle to lateral corner of the eye, base of the nose, labial commissura, and soft tissue pogonion) which was measured with using thread and millimeter ruler.
Postoperative Trismus | Postoperative 2nd day
  Postoperative trismus was evaluated by the maximum distance between the incisive borders of the upper and lower right incisive teeth which was measured with a caliper.
Postoperative Pain | Postoperatif 3th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Pain | Postoperatif 4th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Pain | Postoperatif 5th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Pain | Postoperatif 6th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Pain | Postoperatif 7th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Swelling | Postoperative 7th day
  Postoperative swelling was evaluated by the distance between predetermined facial anatomic landmarks (from the mandibular angle to lateral corner of the eye, base of the nose, labial commissura, and soft tissue pogonion) which was measured with using thread and millimeter ruler.
Postoperative Trismus | Postoperative 7th day
  Postoperative trismus was evaluated by the maximum distance between the incisive borders of the upper and lower right incisive teeth which was measured with a caliper.

CONTACTS AND LOCATIONS:
Overall Officials: Serap KESKIN TUNC, PhD, Study Chair — Cairo University
Locations (1):
- Van Yuzuncu Yil University, Faculty of Dentistry, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No